CLINICAL TRIAL: NCT05907551
Title: Study in Patients With Solid Tumor Regarding Access to Dermo-cosmetics and Aesthetic Solutions
Acronym: DERMOCOS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institut de cancérologie Strasbourg Europe (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-001; 2023-A00546-39 (Other: ID-RCB Number)
Record Dates: First submitted 2023-06-08; First posted 2023-06-18 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Patients with Digestive System Cancer
  Interventions: Other: Questionnaires
- Patients with Head and Neck Cancer
  Interventions: Other: Questionnaires
- Patients with Breast Cancer
  Interventions: Other: Questionnaires
- Patients with Nervous System Tumors
  Interventions: Other: Questionnaires
- Patients with Urological Cancer
  Interventions: Other: Questionnaires
- Patients with Lung Cancer
  Interventions: Other: Questionnaires
- Patients with Gynecologic Cancer
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — 25-items questionnaire

SUMMARY:
Cancer treatments can trigger cutaneous side-effects, as well as nail and hair toxicities. When related to drug treatment, this iatrogeny depends on the type of drug, its dosage and individual susceptibility. Although these dermatological adverse events are rarely serious, they can significantly alter patients' quality of life, and may even necessitate the introduction of curative treatment.

The impact of these side effects can be mitigated by the use of dermo-cosmetic products and aesthetic solutions. However, most of this supportive care is not reimbursed by the health insurance system, representing a source of inequalities in access to healthcare for cancer patients.

DETAILED DESCRIPTION:
This study aims at establishing, in a cohort of patients with solid tumors, the state of their knowledges, given information and their financial capacities regarding access to dermo-cosmetics and aesthetic solutions, that are used in the attenuation of cancer treatments' side-effects.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Patients with solid tumors (eligible localization include: digestive system, Head and Neck, Breast, Brain, Lung Tumors, Urological and Gynecologic cancers)
* Patients able to read and understand French
* Patients that has expressed their consent and with signed consent form

Exclusion Criteria:

* Minor or patients placed under guardianship or supervision
* Patients unable to read French
* Patients placed under judicial protection

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study will enroll patients with solid tumors in 7 different cohorts according to tumor location (30 patients per location)
Sampling Method: Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2023-07-25 (Actual); Primary Completion 2023-10-25 (Estimated); Study Completion 2023-10-25 (Estimated)

PRIMARY OUTCOMES:
Describe patients' knowledges regarding cutaneous side-effects, nail and hair toxicities induced by anticancer drugs | at inclusion
  4 items questionnaires
Describe patients' knowledges regarding dermo-cosmetics and aesthetic solutions that can attenuate cutaneous side-effects, nail and hair toxicities induced by anticancer drugs | at inclusion
  10 items questionnaires

SECONDARY OUTCOMES:
Describe patients' socio-economic profile to assess equity regarding access to dermo-cosmetics and aesthetic solutions | at inclusion
  11 items questionnaires
Correlate patients' knowledge level depending on tumoral location | at inclusion
  Tumoral location as described in medical chart
Correlate patients' knowledge level depending on received treatment | at inclusion
  Type of chemotherapy administered on the day of inclusion as described in medical chart
Correlate patients' knowledge level depending on treatment phase | at inclusion
  Type of treatment phase (i.e. neoadjuvant, adjuvant, 1st or 2nd metastatic line) as described in medical chart

CONTACTS AND LOCATIONS:
Overall Officials: Nelly ETIENNE-SELLOUM, PharmD, Study Chair — Institut de cancérologie Strasbourg Europe
Locations (1):
- Institut de cancérologie Strasbourg Europe, Strasbourg, France